CLINICAL TRIAL: NCT04043416
Title: Using Motivating Reminiscence Technology to Encourage Physical Activity and Improve Balance and Mobility for Residents in Long Term Care
Brief Title: Reminiscence Technology Balance and Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Principal Investigator, Mark Campbell, Clinician-Investigator and Associate Staff Physician, Bruyère Health Research Institute.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M16-19-012
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Results first posted 2020-07-21 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Adults Living in Long Term Care
Keywords: Long Term Care; Motivating Reminiscence Technology; Feasibility

STUDY DESIGN:
Intervention Model Description: This study has 2 six week campaigns with a six week washout in between the 2 campaigns. During the first campaign half of the participants will use the motivating reminiscence technology while receiving the standard fall prevention programming, while the second half will receive just the standard fall prevention programming. During the 6 week washout period all participants will just receive the standard fall prevention programming. After the washout period, there will be the second campaign where the other half of the participants will use the motivating reminiscence technology while receiving the standard fall prevention programming, whereas the remaining participants will just receive the standard fall prevention programming.
Who Masked: Outcomes Assessor
Masking Description: All outcome measures will be collected by the physiotherapy team at The Glebe Centre. The physiotherapy team will be blinded to the group allocation of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- System + Fall Prevention First, then Fall Prevention (Experimental): Participants in this arm will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the first 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program. Following the 6 week washout period, the participants in this arm will just participate in the Fall Prevention program alone.
  Fall Prevention Program focuses on reducing the incidence of residents' falls and mitigating risks of falls through a resident focused, team approach which ensures that a resident's environment and social, physical, cognitive and emotional strengths are supported. This is an interdisciplinary program involving nursing and program staff, physician/pharmacist, dietician, physiotherapist, housekeeping staff and the resident/POA. They communicate regarding their planned interventions and evaluation of resident progress and outcomes in falls prevention through documentation.
  Interventions: Other: Motivating reminiscence technology
- Fall Prevention first, then System +Fall Prevention (Experimental): Participants in this arm will participate in the Fall Prevention program alone during the first 6 week campaign. Following the 6 week washout period the participants will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the second 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program
  Fall Prevention Program focuses on reducing the incidence of residents' falls and mitigating risks of falls through a resident focused, team approach which ensures that a resident's environment and social, physical, cognitive and emotional strengths are supported. This is an interdisciplinary program involving nursing and program staff, physician/pharmacist, dietician, physiotherapist, housekeeping staff and the resident/POA. They communicate regarding their planned interventions and evaluation of resident progress and outcomes in falls prevention through documentation.
  Interventions: Other: Motivating reminiscence technology

INTERVENTIONS:
Other: Motivating reminiscence technology — The jDome BikeAround uses Google Street View, a stationary bike and a domed screen. Residents are seated in front of the screen; their destination is typed into the computer and when loaded the image appears on the screen. Using pedals on the bike they can propel themselves down the street, steer and change direction as they wish.
  Other Names: jDome BikeAround System

SUMMARY:
This study evaluates the feasibility of a larger randomized controlled trial to examine the effect of reminiscence aided physical activity on the balance and mobility of older adults living in long term care. The study uses the jDome BikeAround system, which is a stationary bicycle with a projector screen that runs google earth, as the user bicycles, the map progresses giving the appearance that the user is bicycling through the environment chosen. Half of the participants will use the system during the first 6 week campaign, there will then be a 6 week washout period. Following the washout period, there will be a second 6 week campaign when the other half of the participants will use the jDome BikeAround system.

DETAILED DESCRIPTION:
Physical activity has been shown to have numerous benefits for physical well-being and function. Stationary cycling is one example of physical activity that can provide opportunities for residents who are inactive, living in long term care and are at high risk for falls.

The use of jDome BikeAround provides older adults in long term care an opportunity to engage in a motivating reminiscence activity that is coupled with physical activity. Participants will be divided into two groups, one group will take part in jDome BikeAround sessions 3x per week for 6 weeks in addition to The Glebe Centre's Fall Prevention program, while the second group will just participant in Fall Prevention program. There will be a 6 week wash out, then the second cohort will participant in the jDome Bike Around sessions 3x a week in addition to the Fall Prevention program while the first cohort will just participate in the Fall Prevention Program.

Participants will have their balance, mobility, leg strength, endurance tested as well as a tracking of fall risks at the beginning and end of each of the jDome BikeAround sessions (4 measurement points). Feasibility will be determined by the ability to enroll an adequate number of participants, protocol completion by participants, and the number of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Scott fall risk of 2-17 (this is the current range used by the Glebe Centre, there have been 0 falls during transportation to the equipment and during each session of the BikeAround system)
* Sufficient visual abilities to observe images on the domed screen
* Able to comprehend and communicate in English.
* Adequate attentional capacity to remain focused on the pedalling task.
* Minimum height requirement of 5'2" or 157cm in order to successfully fit the BikeAround system's stationary bike.

Exclusion Criteria:

* Physical limitations (as determined by the Glebe Centre healthcare/physiotherapy team) that prevent use of the jDome bike.
* Cognitive impairment (as determined by the Glebe Centre healthcare/physiotherapy team) Inability to sustain attention Inability to follow one-step commands.
* Known behavioural abnormalities (e.g. overly aggressive behavior) that in the opinion of the clinical care team might impede any meaningful participation in the project
* Those who are in the opinion of attending physician or clinical team too unwell to participate in the project
* Fully unable to complete outcome measures indicated (Section 7, Outcomes)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Campbell, MD, MSc, Principal Investigator — Bruyere Continuing Care
Locations (1):
- The Glebe Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We will not be making IPD available to other researchers.

REFERENCES:
- [Background] Lautenschlager NT, Cox K, Kurz AF. Physical activity and mild cognitive impairment and Alzheimer's disease. Curr Neurol Neurosci Rep. 2010 Sep;10(5):352-8. doi: 10.1007/s11910-010-0121-7. PMID 20556547
- [Background] Vogel T, Brechat PH, Lepretre PM, Kaltenbach G, Berthel M, Lonsdorfer J. Health benefits of physical activity in older patients: a review. Int J Clin Pract. 2009 Feb;63(2):303-20. doi: 10.1111/j.1742-1241.2008.01957.x. PMID 19196369
- [Background] Menne HL, Johnson JD, Whitlatch CJ, Schwartz SM. Activity Preferences of Persons With Dementia. Activities, Adaptation & Aging, 36(3): 195-213, 2012. DOI: 10.1080/01924788.2012.696234
- [Background] Benjamin K, Edwards N, Ploeg J, Legault F. Barriers to physical activity and restorative care for residents in long-term care: a review of the literature. J Aging Phys Act. 2014 Jan;22(1):154-65. doi: 10.1123/japa.2012-0139. Epub 2013 Feb 20. PMID 23434919
- [Background] de Hollander EL, Proper KI. Physical activity levels of adults with various physical disabilities. Prev Med Rep. 2018 Apr 24;10:370-376. doi: 10.1016/j.pmedr.2018.04.017. eCollection 2018 Jun. PMID 29755934
- [Background] Varela S, Cancela JM, Seijo-Martinez M, Ayan C. Self-Paced Cycling Improves Cognition on Institutionalized Older Adults Without Known Cognitive Impairment: A 15-Month Randomized Controlled Trial. J Aging Phys Act. 2018 Oct 1;26(4):614-623. doi: 10.1123/japa.2017-0135. Epub 2018 Sep 8. PMID 29431549
- [Background] Batcir S, Melzer I. Daily Bicycling in Older Adults May be Effective to Reduce Fall Risks-A Case-Control Study. J Aging Phys Act. 2018 Oct 1;26(4):570-576. doi: 10.1123/japa.2017-0263. Epub 2018 Aug 29. PMID 29345533
- [Background] Harvey S, Rissel C, Pijnappels M. Associations Between Bicycling and Reduced Fall-Related Physical Performance in Older Adults. J Aging Phys Act. 2018 Jul 1;26(3):514-519. doi: 10.1123/japa.2017-0243. Epub 2018 Jun 22. PMID 29182418
- [Background] Macaluso A, Young A, Gibb KS, Rowe DA, De Vito G. Cycling as a novel approach to resistance training increases muscle strength, power, and selected functional abilities in healthy older women. J Appl Physiol (1985). 2003 Dec;95(6):2544-53. doi: 10.1152/japplphysiol.00416.2003. Epub 2003 Aug 22. PMID 12937026
- [Background] Huang HC, Chen YT, Chen PY, Huey-Lan Hu S, Liu F, Kuo YL, Chiu HY. Reminiscence Therapy Improves Cognitive Functions and Reduces Depressive Symptoms in Elderly People With Dementia: A Meta-Analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2015 Dec;16(12):1087-94. doi: 10.1016/j.jamda.2015.07.010. Epub 2015 Sep 1. PMID 26341034
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076

RESULTS

PARTICIPANT FLOW:
Groups:
- System+Fall Prevention First, Then Fall Prevention Alone: Participants in this arm will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the first 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program. Following the 6 week washout period, the participants in this arm will just participate in the Fall Prevention program alone.
  Fall Prevention Program focuses on reducing the incidence of residents' falls and mitigating risks of falls through a resident focused, team approach which ensures that a resident's environment and social, physical, cognitive and emotional strengths are supported. This is an interdisciplinary program involving nursing and program staff, physician/pharmacist, dietician, physiotherapist, housekeeping staff and the resident/POA. They communicate regarding their planned interventions and evaluation of resident progress and outcomes in falls prevention through documentation.
- Fall Prevention First, Then System+Fall Prevention: Participants in this arm will participate in the Fall Prevention program alone during the first 6 week campaign. Following the 6 week washout period the participants will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the second 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program Fall Prevention Program focuses on reducing the incidence of residents' falls and mitigating risks of falls through a resident focused, team approach which ensures that a resident's environment and social, physical, cognitive and emotional strengths are supported. This is an interdisciplinary program involving nursing and program staff, physician/pharmacist, dietician, physiotherapist, housekeeping staff and the resident/POA. They communicate regarding their planned interventions and evaluation of resident progress and outcomes in falls prevention through documentation.
Period: Campaign 1
Arm/Group | System+Fall Prevention First, Then Fall Prevention Alone | Fall Prevention First, Then System+Fall Prevention
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout
Arm/Group | System+Fall Prevention First, Then Fall Prevention Alone | Fall Prevention First, Then System+Fall Prevention
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1
Not completed — Change in health condition | 0 | 1
Period: Campaign 2
Arm/Group | System+Fall Prevention First, Then Fall Prevention Alone | Fall Prevention First, Then System+Fall Prevention
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant who was part of the cohort using the campaign during the second campaign was withdrawn from the study due to an injury that occurred during the washout period between the two campaigns. This injury was not study related.
Groups:
- System + Fall Prevention First, Then Fall Prevention: Participants in this arm will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the first 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program. Following the 6 week washout period, the participants in this arm will just participate in the Fall Prevention program alone.
  Motivating reminiscence technology: The jDome BikeAround uses Google Street V
- Fall Prevention First, Then System +Fall Prevention: Participants in this arm will participate in the Fall Prevention program alone during the first 6 week campaign. Following the 6 week washout period the participants will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the second 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program
  Motivating reminiscence technology: The jDome BikeAround uses Google Street V
- Total: Total of all reporting groups
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 87.7 (9.9) | 79.9 (9.1) | 84.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 13 | 27
Scott Fall Risk [Mean (Standard Deviation); unit: units on a scale] — Scott Fall Risk is an assessment tool that measures the risk of falls for a resident in long term care. The higher the value on the assessment indicates a higher risk of falls and the range is -5 - 19. A score below 7 indicates that universal fall precautions with a plan for individual risks need to be in place for that individual, a score equal to or greater than 7 but equal to or less than 12 indicates the individual is at high risk for a fall and a score above 12 indicates the individual is at a high risk for a fall and has unsafe ambulation.
  units on a scale | 7.1 (4.7) | 8.9 (5.3) | 8.0 (5.0)
Cognitive Performance Scale (CPS) [Mean (Standard Deviation); unit: units on a scale] — CPS is tool to assess the cognitive abilities of residents living in long-term care. CPS has a range 0-5, the higher the value the greater the cognitive impairment
  units on a scale | 3 (0.8) | 3 (1.3) | 3 (1.1)
Index for Social Engagement (ISE) [Mean (Standard Deviation); unit: units on a scale] — Index for Social Engagement assess a resident's social engagement while living in Long Term Care. The range is 0-6 and a higher scores indicate a higher level of social engagement
  units on a scale | 5 (1.3) | 5 (1.2) | 5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: Determine the feasibility of a future randomized controlled trial to evaluate the impact on balance and mobility of motivating reminiscence technology using the jDome BikeAround system for adults in long term care. Feasibility will be determined by the ability to recruit 30 residents (based on the LTC population base at The Glebe Centre).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 14 | 14
Participants | 14 | 14

2. Primary Outcome: Protocol Adherence
Description: Determine the feasibility of a future randomized controlled trial to evaluate the impact on balance and mobility of motivating reminiscence technology using the jDome BikeAround system for adults in long term care. Feasibility will be determined by the number of residents to complied with the protocol during their respective campaign by using the jDome BikeAround system 3 times a week.
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 14 | 13
Participants | 2 | 4

3. Primary Outcome: Number of Participants Who Experience an Adverse Events While Using the jDome BikeAround (System)
Description: The number of adverse events while directly interacting with the jDome BikeAround system will be tracked to help determine feasibility of this kind of randomized trial.
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 14 | 13
Participants | 0 | 0

4. Primary Outcome: Performance Oriented Mobility Assessment
Description: The Performance Oriented Mobility Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks as either 0, 1 or 2 where a score of 0 represents the most impaired while a score of 2 represents independence. The total is calculated by adding the score for each individual activity, the lowest possible score is 0 and the highest possible score is 28. The higher the score the better the more mobile the participant is. This will give us a baseline value for the participants.
Time Frame: Baseline
Population: To complete this test, the participant must have a certain level of mobility. Out of the 14 participants in the "System + Fall Prevention First, then Fall Prevention" cohort, 4 couldn't complete the test.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- System + Fall Prevention First, Then Fall Prevention: Participants in this arm will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the first 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program. Following the 6 week washout period, the participants in this arm will just participate in the Fall Prevention program alone.
  Motivating reminiscence technology: The jDome BikeAround
- Fall Prevention First, Then System +Fall Prevention: Participants in this arm will participate in the Fall Prevention program alone during the first 6 week campaign. Following the 6 week washout period the participants will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the second 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 10 | 14
units on a scale | 19.6 (2.9) | 21.6 (3.7)

5. Primary Outcome: Performance Oriented Mobility Assessment
Description: The Performance Oriented Mobility Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks as either 0, 1 or 2 where a score of 0 represents the most impaired while a score of 2 represents independence. The total is calculated by adding the score for each individual activity, the lowest possible score is 0 and the highest possible score is 28. The higher the score the better the more mobile the participant is. This measure will be taken after the first campaign has been completed.
Time Frame: Week 6
Population: To complete this test, the participant must have a certain level of mobility. Out of the 14 participants in the "Motivating reminiscence technology + Fall Prevention" cohort, 3 couldn't complete the test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 11 | 13
units on a scale | 16.8 (6.5) | 19.6 (6.7)

6. Primary Outcome: Performance Oriented Mobility Assessment
Description: The Performance Oriented Mobility Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks as either 0, 1 or 2 where a score of 0 represents the most impaired while a score of 2 represents independence. The total is calculated by adding the score for each individual activity, the lowest possible score is 0 and the highest possible score is 28. The higher the score the better the more mobile the participant is. This measure will be taken just before the second campaign is to begin.
Time Frame: Week 12
Population: To complete this test, the participant must have a certain level of mobility. Out of the 14 participants in the "System + Fall Prevention First, then Fall Prevention" cohort, 5 couldn't complete the test and 2 participant out of the 13 participants in the 'Fall Prevention first, then System +Fall Prevention' cohort that could not complete the test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 9 | 11
units on a scale | 16.5 (7.6) | 19.7 (7.6)

7. Primary Outcome: Performance Oriented Mobility Assessment
Description: The Performance Oriented Mobility Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks as either 0, 1 or 2 where a score of 0 represents the most impaired while a score of 2 represents independence. The total is calculated by adding the score for each individual activity, the lowest possible score is 0 and the highest possible score is 28. The higher the score the better the more mobile the participant is. This measure will be taken after the second campaign has been completed.
Time Frame: Week 18
Population: To complete this test, the participant must have a certain level of mobility. Out of the 14 participants in the "System + Fall Prevention First, then Fall Prevention" cohort, 5 couldn't complete the test and 1 participant out of the 13 in the 'Fall Prevention first, then System +Fall Prevention' cohort that could not complete the test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 9 | 12
units on a scale | 17 (6.8) | 19 (7.6)

8. Secondary Outcome: 2 Minute Walk Test
Description: Distance participant can walk without assistance for 2 minutes measured from the starting position.
Time Frame: Baseline
Population: Due to the inability to ambulate for 2 minutes independently, in the arm "System + Fall Prevention First, then Fall Prevention" 4 residents were unable to complete the test and 2 residents in the "Fall Prevention first, then System +Fall Prevention" were unable to complete the test.
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 10 | 12
Meter | 60.9 (26.5) | 84.7 (55.1)

9. Secondary Outcome: 2 Minute Walk Test
Description: Distance participant can walk without assistance for 2 minutes measured from the starting position.
Time Frame: 6 Week
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Meter
Groups:
- System + Fall Prevention First, Then Fall Prevention: Participants in this arm will be invited to use the jDome BikeAround system for up to 30 minute sessions up to 3 times a week during the first 6 week campaign. During this campaign the participants will also participant in the standard fall prevention program. Following the 6 week washout period, the participants in this arm will just participate in the Fall Prevention program alone.
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 10 | 12
Meter | 72.4 (9.1) | 67.6 (27.1)

10. Secondary Outcome: 2 Minute Walk Test
Description: Distance participant can walk without assistance for 2 minutes measured from the starting position.
Time Frame: 12 Week
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 10 | 11
Meter | 70.7 (27.1) | 68.6 (31.8)

11. Secondary Outcome: 2 Minute Walk Test
Description: Distance participant can walk without assistance for 2 minutes measured from the starting position.
Time Frame: 18 Week
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 10 | 11
Meter | 54.5 (32.5) | 67.6 (27.1)

12. Secondary Outcome: Knee Range of Motion Test
Description: Test that asses the range of motion of a participant's knee
Time Frame: Baseline
Population: 2 participants in the "Fall Prevention first, then System +Fall Prevention" could not have their knee range of motion measures.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 14 | 12
Degrees
  Left Knee Extension | -3.2 (5.8) | -2.9 (4.3)
  Right Knee Extension | -3.6 (8.5) | -2.7 (4.2)
  Left Knee Flexion | 111.6 (12.4) | 109.3 (12.6)
  Right Knee Flexion | 107.2 (17.8) | 106.1 (13.7)

13. Secondary Outcome: Knee Range of Motion Test
Description: Test that asses the range of motion of a participant's knee
Time Frame: 6 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 14 | 12
Degrees
  Left Knee Extension | -1.4 (5.3) | -5 (8.5)
  Right Knee Extension | -2.1 (8.0) | -4.2 (7.6)
  Left Knee Flexion | 114.6 (16.6) | 115.0 (9.5)
  Right Knee Flexion | 115.7 (14.7) | 116.7 (9.8)

14. Secondary Outcome: Knee Range of Motion Test
Description: Test that asses the range of motion of a participant's knee
Time Frame: 12 weeks
Population: One participants in the "System + Fall Prevention First, then Fall Prevention" could not have their knee range of motion measures.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 13 | 13
Degrees
  Left Knee Extension | 0 (6.9) | -1.25 (4.3)
  Right Knee Extension | -2.3 (8.3) | -1.7 (5.8)
  Left Knee Flexion | 118.8 (11.0) | 116.5 (15.7)
  Right Knee Flexion | 116.5 (13.8) | 116.7 (16.3)

15. Secondary Outcome: Knee Range of Motion Test
Description: Test that asses the range of motion of a participant's knee
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
Number analyzed (Participants) | 14 | 13
Degrees
  Left Knee Extension | 0 (0) | 0 (0)
  Right Knee Extension | -0.7 (2.7) | -3.5 (7.7)
  Left Knee Flexion | 110.4 (13.4) | 111.9 (10.7)
  Right Knee Flexion | 111.4 (11.3) | 108.8 (11.2)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | System + Fall Prevention First, Then Fall Prevention | Fall Prevention First, Then System +Fall Prevention
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04043416/Prot_SAP_001.pdf